CLINICAL TRIAL: NCT05925998
Title: Mitochondrial Function in the Peri-operative Setting: an Observational Study
Acronym: MITOSIS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CRI0430
Record Dates: First submitted 2023-06-01; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Mitochondrial; Perioperative Complication; Surgery-Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skeletal muscle, blood plasma/serum, red blood cells, exhaled breath
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study: no interventions — Not applicable as observational study with no intervention

SUMMARY:
Complications after surgery are common and a burden for patients and health services. Therefore it is important that clinicians improve surgical outcomes. Mitochondria are the part of the body's cells that manage energy. Research has already shown that how our body's mitochondria behave can predict who survives in intensive care patients. The investigators think this could also predict who is more likely to develop complications after surgery. Therefore a study has been designed to find out if changes in mitochondria are related to postoperative complications. This will help doctors improve how they prepare patients for surgery and potentially how they manage their treatment, and result in improving outcomes for patients after surgery.

This study will recruit patients scheduled for major abdominal surgery as part of their treatment. The investigators will take samples of breath, blood and muscle to measure changes in mitochondria from the day before surgery to 7 days postoperatively. The muscle samples will only be taken when the patient is asleep having their operation. These samples will be used to analyse mitochondria. This study will be in two phases. Phase 1 is a pilot of up to 10 patients focussed on feasibility. Following this there will be an interim data analysis. The results may allow further optimisation to reduce the patient burden, eg reduction in sampling frequency, or avoiding need for muscle biopsy. The second phase will be a full cohort study of up to 40 patients, focussed on association of mitochondrial markers with clinical outcomes, such as postoperative complications, oxygen levels, pain, confusion and length of intensive care stay.

The results of this study could improve how doctors select and prepare patients for surgery. It may also affect how doctors manage their treatment during and after operations. This could result in reducing complications and illness burden for patients after surgery.

DETAILED DESCRIPTION:
Postoperative mortality is the third highest cause of death globally. Postoperative morbidity is up to 17 times higher than mortality. As well as being a burden for patients, postoperative complications result in excess costs of tens of thousands of dollars (USA) per patient. Complications are also strongly correlated with overall cost in European studies. Increasing evidence suggests that common but essential parts of general anaesthetic techniques, such as administration of supplemental oxygen, may be related to these postoperative outcomes. Work from our group has shown that changes in mitochondrial activity are central to altered oxygen handling seen at high altitude and indirectly suggested this may change during major abdominal surgery. Changes in mitochondrial activity have also already been shown to be distinct between survivors and non-survivors in critical care cohorts. Early unpublished data has also shown there may be some change in mitochondrial signal in skeletal muscle in surgical patients at end of surgery with an average of around 6 hours duration. Therefore, our hypothesis is that mitochondrial function/ activity changes during and in recovery from major abdominal surgery in trajectories associated with different rates of postoperative complications. Establishing this may enable us to predict patient susceptibility to postoperative complications. This would be extremely powerful to enable optimisation of patient selection, preparation and prognostication. It may also lead to changes in intra- and postoperative management. All of these factors could reduce postoperative complications and their associated morbidity and mortality.

A two-stage prospective observational cohort study has been designed to test this hypothesis. The first phase will be a pilot, including up to 10 adult patients scheduled for elective major open abdominal surgery, requiring siting of arterial and central venous lines and admission the day before surgery. This will focus on examining the feasibility of performing multi-modal mitochondrial analysis in surgical patients and charting the trajectory of change in mitochondrial markers through the perioperative period. Blood will be taken around the start of surgery and on postoperative days 1 and 7. Muscle biopsies will be taken around the start of surgery and at end of surgery or 12 hours after start, whichever is soonest. Exhaled breath samples will be taken the day before surgery and on postoperative day 7. High-resolution respirometry will be used for skeletal muscle and platelet analysis ex-vivo with saturating quantities of substrate and oxygen. 13C-ketoisocaproate (13C-KICA) breath tests (BT) will be carried out to measure hepatic and skeletal muscle mitochondrial function representing in-vivo substrate concentrations and intercurrent oxygenation levels. Clinical data and results of routine blood tests and blood gas analysis will also be collected.

Following the pilot phase of up to 10 patients there will be an interim data analysis. This is to allow optimisation of the process following the feasibility phase. It may also provide the opportunity to reduce sampling burden for the patient. For example if it is established that either fewer sampling points are needed, or if muscle and platelet respirometry data correlate it may be possible to remove the need for muscle biopsy in the second phase.

The second phase will include a cohort of up to 40 patients recruited in the same manner and sampled in the same scheme as the pilot, unless it has been possible to reduce the sample burden as a result of the pilot phase data. This phase will aim to establish if changes in mitochondrial activity are related to clinical outcomes.

The primary objective of the pilot phase is: To examine the feasibility of multi-modal mitochondrial analysis in patients undergoing major elective abdominal surgery. This will include the number of eligible patients screened and consented, the optimisation of sampling timepoints and clinical data collection.

Secondary objectives will include:

* Establishing if and how mitochondrial activity measured in platelets and in skeletal muscle relates to each other in surgical patients.
* Relation of postoperative complication rate as measured by day 7 Postoperative Morbidity Survey (POMS), to change in platelet mitochondrial activity from start of surgery to day 1 postoperatively, as measured by high resolution respirometry.
* Description of the trajectories of change in respiratory capacity/ mitochondrial function through the perioperative period as measured by respirometry in platelets and skeletal muscle, and by 13C-KICA breath test.
* Relation of postoperative complication rate to change in skeletal muscle mitochondrial activity and respiratory capacity, as measured by high resolution respirometry, from start of surgery to 12 hours into surgery/ end of surgery.
* Relation of postoperative complication rate to change in platelet mitochondrial activity and respiratory capacity, as measured by high resolution respirometry, from start of surgery to 7 days postoperatively.
* Relation of postoperative complication rate to change in hepatic and skeletal muscle mitochondrial function as measured by 13C-KICA breath test from baseline to 7 days postoperatively.
* Change in the following criteria in relation to mitochondrial function/ activity as measured by any of the above:

  * Oxygenation parameters (eg. Fraction of inspired oxygen (FiO2), Partial pressure of oxygen in arterial blood (PaO2))
  * Length of stay in ICU/HDU environment prior to ward step-down
  * Duration of postoperative invasive mechanical ventilation
  * Postoperative delirium on day 7 as measured by Confusion Assessment Method (CAM) score
  * Patient reported postoperative pain (score out of 10)
  * Charleston Comorbidity Index

Following the pilot phase of up to 10 patients there will be an interim data analysis. This is to allow optimisation of the process following the feasibility phase. It may also provide the opportunity to reduce sampling burden for the patient. For example if it is established that either fewer sampling points are needed, or if muscle and platelet respirometry data correlate it may be possible to remove the need for muscle biopsy in the second phase.

The second phase will include a cohort of up to 40 patients recruited in the same manner and sampled in the same scheme as the pilot, unless it has been possible to reduce the sample burden as a result of the pilot phase data. This phase will aim to establish if changes in mitochondrial activity are related to clinical outcomes.

The primary objective of the second phase is: to establish any relation of postoperative complication rate as measured by day 7 Postoperative Morbidity Survey (POMS), to change in mitochondrial activity through the perioperative period, as measured by high resolution respirometry.

The secondary objectives will include a subset of those of the pilot phase, established following the interim analysis.

Blood/ muscle/ breath sampling and data collection will be performed by Good Clinical Practice (GCP) -trained researchers or members of the treating clinical team. The definition of the study end is once all analysis has been completed on the final sample. We anticipate the results of this study will be disseminated by publication in a peer-reviewed journal and through conference presentations. Published results will be made available to participants on request.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above.
* Having elective major abdominal surgery under general anaesthesia requiring a CVC and arterial line.
* Planned for a Total Intravenous Anaesthesia (TIVA) technique +/- additional regional or neuraxial anaesthesia.
* Admitted >6 hours prior to planned start of surgery as part of their normal care
* Willingness to donate blood and breath samples to the study; declining muscle biopsy would not preclude inclusion.

Exclusion Criteria:

* Currently pregnant or up to 6 weeks post-partum
* Participating in an interventional research study concerning intra-operative management already
* Lacks capacity to give consent to participate in the study at time of recruitment
* Currently in custody
* Surgery in the past 28 days
* Existing primary mitochondrial disease as defined by previous genetic testing/ genome- or exome- sequencing results, or formal diagnosis by a medical professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults having major elective abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-05 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of eligible patients screened | Through study completion, an average of 3 years
  Number of eligible patients screened
Number of eligible patients consented | Through study completion, an average of 3 years
  Number of eligible patients consented
Postoperative Morbidity Survey (POMS) on day 7 postoperatively | From start of surgery to day 7 postoperatively
  Postoperative Morbidity Survey (POMS) on day 7 postoperatively

SECONDARY OUTCOMES:
Difference in mitochondrial activity in platelets as measured by high resolution respirometry from start of surgery to day 7 postoperatively | From start of surgery to day 7 post-operatively
  Difference in mitochondrial activity in platelets as measured by high resolution respirometry from start of surgery to day 7 postoperatively
Difference in mitochondrial function as measured by 13C-KICA breath test from day before surgery to day 7 postoperatively | From day before surgery to day 7 post-operatively
  Difference in mitochondrial function as measured by 13C-KICA breath test from day before surgery to day 7 postoperatively
Difference in mitochondrial activity in skeletal muscle as measured by high resolution respirometry from start of surgery to day 1 postoperatively | From start of surgery to day 1 post-operatively
  Difference in mitochondrial activity in skeletal muscle as measured by high resolution respirometry from start of surgery to day 1 postoperatively
Length of stay in ICU/HDU environment prior to ward step-down | From start of surgery to day 7 post-operatively
  Length of stay in ICU/HDU environment prior to ward step-down
Duration of postoperative invasive mechanical ventilation | From start of surgery to day 7 post-operatively
  Duration of postoperative invasive mechanical ventilation
Charleston Comorbidity Index on postoperative days 3,4,5 and 7 | From start of surgery to day 7 post-operatively
  Charleston Comorbidity Index on postoperative days 3,4,5 and 7

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
If participants consent (written) to their data being shared, their anonymised data such as laboratory results may be shared with other researchers.